CLINICAL TRIAL: NCT07008963
Title: A Non-interventional, Observational Qualitative Interview Study of Patients With HR+/HER2- Metastatic Breast Cancer Who Received Capivasertib + Fulvestrant
Brief Title: Interview of Patients With HR+/HER2- Metastatic Breast Cancer Who Received Capivasertib + Fulvestrant
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3615R00004
Record Dates: First submitted 2025-05-05; First posted 2025-06-06 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes

INTERVENTIONS:
Other: non-interventional — This is a non-interventional, observational study

SUMMARY:
A cross-sectional, non-interventional, observational study using qualitative patient interviews to explore patient experiences and attitudes toward taking capivasertib + fulvestrant as directed

ELIGIBILITY:
Inclusion criteria (self-reported):

* Adult (over the age of 18 years)
* Diagnosed with HR+/HER2- metastatic breast cancer
* Received at least 1 week of capivasertib + fulvestrant (Patients will be invited to provide documents demonstrating the use of capivasertib. Patients will be able to participate even if unable to obtain such documentation)

Exclusion criteria (self-reported):

* Patients who had discontinued capivasertib for more than 6 months before the date of the interview
* Unable or unwilling to follow study procedures (including providing informed consent)
* Not proficient in spoken English, as assessed by the moderator
* Receiving capivasertib in a clinical trial setting
* Patients who are not able to recall instruction for administration of capivasertib in a manner consistent with the labeling (e.g. 4 days on followed by 3 days off)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults patients with HR+/HER2- metastatic breast cancer who received capivasertib + fulvestrant
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient attitude and experience reported by patients regarding capivasertib dosing schedule and regimen | Day 1
  The interview will be conducted using a discussion guide tailored to specific questions to be explored in this study, developed by the study team. No formal scale or validated questionnaire will be used to assess the outcomes

SECONDARY OUTCOMES:
Self-reported tolerability experiences related to patients' ability to follow the prescribed regimen and stay on treatment among those who received capivasertib + fulvestrant. | Day 1
  The interview will be conducted using a discussion guide tailored to specific questions to be explored in this study, developed by the study team. No formal scale or validated questionnaire will be used to assess the outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Redwood Shores, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/